CLINICAL TRIAL: NCT07036731
Title: A Prospective, Multicenter, Randomized Study Comparing the Necessity of a Second Transurethral Resection in High-Risk Non-Muscle-Invasive Bladder Cancer Patients With Negative Results From Post-Initial Resection Urine Genome-Wide Low-Depth Sequencing
Brief Title: A Study Comparing the Necessity of a Second Transurethral Resection in High-Risk Non-Muscle-Invasive Bladder Cancer Patients With Negative Results From Post-Initial Resection Urine Genome-Wide Low-Depth Sequencing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Qiang Lv, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-310
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: reTURBT; NMIBC; urine biomarker; RFS
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Fanconi Syndrome

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria are randomized 1:2 into two parallel groups. Group A: Participants assigned to this group will not undergo reTURBT. They will receive standard follow-up care as per institutional guidelines.
  Group B: Participants assigned to this group will undergo reTURBT as part of their treatment protocol. Following reTURBT, they will also receive standard follow-up care. Outcome measures of recurrence rate and RFS would be compared between the two groups to determine the effectiveness and safety of the urine genetic test-guided approach compared to standard care with reTURBT.Throughout the study period, both groups are followed up simultaneously, allowing for parallel comparisons of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine biomarker -Guided without reTURBT (Experimental): Participants in this arm will proceed without reTURBT if Urine biomarker tested negative
  Interventions: Procedure: Urine biomarker -Guided without reTURBT
- Standard Care with reTURBT (No Intervention): Participants in this arm will receive standard care, which undergo reTURBT

INTERVENTIONS:
Procedure: Urine biomarker -Guided without reTURBT — Participants will proceed without reTURBT
  Arms: Urine biomarker -Guided without reTURBT

SUMMARY:
This study is a prospective, randomized, multicenter clinical trial aiming to enroll 428 patients with non-muscle-invasive bladder cancer (NMIBC) from the Department of Urology at Jiangsu Provincial People's Hospital and its affiliated centers, who have undergone their initial transurethral resection and are scheduled for a second resection. Within 1-6 weeks after the first resection and prior to the second resection, 100ml of routine urine will be collected and sent within 24 hours to Beijing Genetron Health Clinical Laboratory Co., Ltd. for the extraction of urinary sediment DNA, which will then undergo genome-wide low-depth sequencing. Patients with positive test results will proceed with the second resection, while those with negative results will be randomly assigned in a 1:2 ratio to either the intervention group, which will not undergo a second resection, or the control group, which will undergo the second resection. All enrolled patients will be followed up for two years. The study will statistically analyze and compare the two-year recurrence-free survival rates between the two groups and evaluate the predictive capability of the test results for follow-up recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NMIBC who have completed the initial transurethral resection and are scheduled for a second resection, as recommended by guidelines or physician's choice:

  1. Incomplete initial TURBT due to various reasons (including large tumor size, high risk of intraoperative bleeding, extensive tumor range, etc.), posing a risk of residual tumor;
  2. Absence of muscle layer tissue in the initial resection specimen;
  3. Post-initial resection pathology indicating T1 stage;
  4. Post-initial resection pathology indicating G3/high-grade tumor, excluding pure carcinoma in situ;
* Ability to provide a 100ml routine urine sample within 1-6 weeks after the initial resection and before the second resection;
* Age ≥ 18 years;
* Willingness to provide basic clinical information, pathology, and subsequent - recurrence monitoring results;
* Willingness to sign the informed consent form.

Exclusion Criteria:

* Patients with other non-urothelial malignant tumors (including prostate cancer and renal cell carcinoma);
* Patients previously diagnosed with muscle-invasive bladder cancer;
* Patients unable to undergo a second resection;
* Patients with incomplete pathological information of the sample;
* Patients with contaminated samples;
* Patients whose urine samples fail quality control for valid reasons and cannot be resampled;
* Any condition deemed by the investigator as potentially harming the subject or preventing the subject from meeting or fulfilling the study requirements;
* Patients unable to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
2-year RFS rate | from initial TURBT to the first confirmed recurrence within 2 years
  the proportion of participants experiencing a recurrence during follow-up within 2 years

SECONDARY OUTCOMES:
RFS | from initial TURBT to the first confirmed recurrence within 2 years
  the duration from the completion of initial TURBT until the first recurrence of cancer is detected or until the end of the follow-up period, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu 210029, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR